CLINICAL TRIAL: NCT02225067
Title: Unblinded Comparison Study for Relationship and Reproducibility Between C13-CAC Breath Test and 24-hour Gastric pH Monitoring, in Patients With Acid-related Diseases and Healthy Volunteers
Brief Title: Comparison Study Between C13-CAC Breath Test and 24-hour Gastric pH Monitoring
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: EPS Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAC-14-001
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Acid-related Diseases; Healthy
Keywords: Patients; Volunteers
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C13-CAC (Experimental)
  Interventions: Drug: Calcium (13C)Carbonate

INTERVENTIONS:
Drug: Calcium (13C)Carbonate — Visit 1 and Visit 2, 24-hour gastric pH monitoring and C13-CAC breath test containing 200 mg of Calcium (13C)Carbonate

SUMMARY:
The purpose of this study is to compare C13-CAC Breath Test with 24-hour Gastric pH Monitoring in Patients with Gastric Acid-related Diseases and Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gastric Acid-related diseases like peptic ulcer or gastroesophageal reflux disease in investigator's judgment
* Healthy subjects who are determined no history of Helicobacter pylori infections

Exclusion Criteria:

* Patients with hypercalcemia
* Patients with hypothyroidism
* Patients with hyperparathyroidism
* History of upper gastrointestinal surgery or resection
* Any condition would limit the subject's ability to complete 24-hour gastric pH monitoring

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
13CO2 concentration in expired air | 5，10，15，20，25，30，40，50，60，80，100 and 120minutes after C13-CAC administration
  13CO2 concentration in expired air, 13CO2 excretion rate in expired air as well as the pharmacokinetic parameters (Cmax, AUCt, AUC∞, tmax, λz, and t1/2) determined from the 13CO2 concentration in expired air and 13CO2 excretion rate in expired air
24-hour gastric pH | from completion of pre-study examination to before C13-CAC adminitration
  Gastric pH immediately before taking the C13-CAC and mean gastric pH from a specified time point to the time before C13-CAC administration

OTHER OUTCOMES:
Gastric pH holding time ratio | from completion of pre-study examination to before C13-CAC adminitration
  pH 3 holding time ratio and pH 4 holding time ratio in the 24-hour gastric pH monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Kimiyoshi Sudoh, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- OPHAC Hospital, Osaka, Osaka, Japan